CLINICAL TRIAL: NCT06360549
Title: Effect of Percutaneous Acupoint Electrical Stimulation on Delirium After Thoracoscopic Pneumonectomy
Brief Title: Effect of Percutaneous Acupoint Electrical Stimulation on Delirium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qin Zhang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-IRB202403019
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Delirium, Postoperative
Keywords: Delirium; Thoracoscopic lung resection surgery
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: The intervention group was percutaneous acupoint electrical stimulation treatment group, and the control group was conventional treatment group.
  Inclusion criteria:
  1. Voluntarily sign informed consent;
  2. Age ≥18 years old;
  3. Patients undergoing thoracoscopic pneumonectomy;
  4. ASA Grade I-III;
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (No Intervention): • Intrabronchial general anesthesia was used for anesthesia in all patients. Electrocardiogram (ECG), pulse oxygen saturation (SpO2), blood pressure (BP), body temperature (T), end-expiratory carbon dioxide (EtCO2), ventilators related parameters (VT, f, MV, etc.), and EEG monitoring (BIS) were routinely monitored during the operation.
- Percutaneous acupoint electrical stimulation treatment group (Experimental): On the basis of the conventional treatment received by the control group, the following additional treatments were implemented: Patients assigned to the treatment group underwent acupuncture with electrode pieces placed on bilateral Sanyin jiao, bilateral Zusanli, bilateral Shenmen, Shenting, Yintang, bilateral Hegu, and bilateral Neiguan 30 minutes before anesthesia. The acupuncture involved electrical stimulation using a dense wave with a frequency of 2/100Hz. The stimulation intensity was adjusted to the maximum current tolerable by the patient, typically ranging from 1-7mA, and continued until the conclusion of the operation.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Acupoint Stimulation — Transcutaneous Electrical Acupoint Stimulation (TEAS) is a treatment that combines acupoint theory of traditional Chinese medicine with modern electrical stimulation techniques. It achieves the purpose of acupoint stimulation by applying a weak current to a specific part. TEAS operate just like ordinary electrodes with non-invasive, safe, portable, adjustable and other advantages.
  Arms: Percutaneous acupoint electrical stimulation treatment group

SUMMARY:
This study is a multicenter, prospective, randomized controlled clinical trial that aims to observe the impact of Transcutaneous Electrical Acupoint Stimulation (TEAS) on plasma TK/MMP3 in a randomized controlled setting. The intervention group received percutaneous acupoint electrical stimulation, whereas the control group underwent conventional treatment. The primary objective is to enhance the management of postoperative delirium, specifically focusing on the occurrence and severity of delirium following thoracoscopic pulmonary resection. Additionally, various perioperative inflammatory markers, cognitive function, recovery quality, pain levels, anxiety, sleep patterns, postoperative complications, and overall hospital stay duration were monitored to elucidate the mechanisms through which percutaneous acupoint electrical stimulation improves postoperative delirium.

DETAILED DESCRIPTION:
Transcutaneous Electrical Acupoint Stimulation (TEAS) is a treatment method that combines acupuncture point theory of traditional Chinese medicine with physical electrical stimulation techniques. It achieves the purpose of acupoint stimulation by applying a weak current to a specific part. Compared with traditional acupuncture, TEAS has the advantages of non-invasiveness, safety, portability and adjustability. Intraoperative acupoint electrical stimulation has no effect on operation and monitoring.

This multicenter, prospective, randomized controlled clinical trial aims to investigate the impact of Transcutaneous Electrical Acupoint Stimulation (TEAS) on postoperative delirium following thoracoscopic pulmonary resection. The study design involves the randomized allocation of participants into two groups: an intervention group receiving percutaneous acupoint electrical stimulation and a control group undergoing standard postoperative care.

The intervention protocol includes the precise selection of acupoints for TEAS application, parameters for electrical stimulation, frequency of treatments, and duration of intervention sessions. Patients in the control group will receive conventional postoperative management without TEAS.

Outcome measures will assess plasma TK/MMP3 levels, incidence and severity of postoperative delirium, perioperative inflammatory markers, cognitive function, pain levels, anxiety, sleep patterns, postoperative complications, recovery quality, and hospital stay duration. Statistical analysis will employ appropriate methods to evaluate the effectiveness of TEAS in managing postoperative delirium.

Overall, this clinical trial seeks to contribute to the understanding of how TEAS may improve postoperative delirium management and patient outcomes following thoracoscopic pulmonary resection. The Detailed Description provides a comprehensive overview of the study protocol without duplicating information presented elsewhere in the document.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study;
* Age ≥ 18 years;
* Patients scheduled for thoracoscopic lung resection surgery;
* ASA grade I-III.

Exclusion Criteria:

* History of severe central nervous system diseases, psychiatric disorders, cognitive impairment, intellectual disability, or Mini-Mental State Examination (MMSE) score ≤23;
* History of opioid addiction, long-term use of analgesic drugs, or psychotropic drugs;
* Severe cardiovascular and cerebrovascular diseases;
* Severe liver and kidney dysfunction: Child-Pugh grade B, C patients, patients requiring regular dialysis, etc.;
* Pregnant or postpartum women;
* Patients with language communication barriers;
* Deemed unsuitable for participation by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Delirium (using the Delirium Rating Scale, DRS) | Recovery period, 24 hours after surgery, 72 hours after surgery, 7 days after surgery
  The Delirium Rating Scale (DRS) is a validated instrument used to assess the severity of delirium in individuals. The DRS total score ranges from 0 to 46, with higher scores indicating greater severity of delirium symptoms.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Recovery period, 24 hours after surgery, 72 hours after surgery, 7 days after surgery
  The Mini-Mental State Examination (MMSE) is a widely used cognitive screening tool that assesses various cognitive functions, including orientation, memory, attention, and language. The total score ranges from 0 to 30, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, phd, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei